CLINICAL TRIAL: NCT05649592
Title: Imaging Characteristics of Chronic Lumbar Disc Herniation From the Perspective of Core Muscles and Subcutaneous Fat Tissue Thickness: an Observational Study
Brief Title: Imaging Characteristics of Chronic Lumbar Disc Herniation From the Perspective of Core Muscles and Subcutaneous Fat Tissue Thickness
Acronym: ICCLDHPCMSFT
Status: Completed | Type: Observational
Sponsor: Zhan Yunfan (Other)
Responsible Party: Sponsor-Investigator, Zhan Yunfan, ShuGuang Hospita, ShuGuang Hospital
Organization: ShuGuang Hospital (Other)
Other Study IDs: 3568185739
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Lumbar disc herniation patients
  Interventions: Diagnostic Test: Magnetic Resonance Hydrolipid Separation Imaging
- healthy volunteers
  Interventions: Diagnostic Test: Magnetic Resonance Hydrolipid Separation Imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Hydrolipid Separation Imaging — MRHS was used to measure different muscle percent fat of core muscles. MRHS, also called Dixon imaging, mainly used the different resonant frequency between the hydrogen nuclei in water and in fat to perform the data acquisition at different echo times (TE). The Dixon sequence basically acquires two images, one image with water and fat signals in-phase and the other with water and fat signals out-of-phase: the sum and subtraction of the two images allow the production of a water-only image and a fat-only image. Scanning equipment: 3.0T superconducting Siemens Skyra Scanner.
  Scanning parameters: TR5.36ms, TE1.24ms, Flip Angle 9°, number of layers was 44-60, thickness of layer was 5.0 mm, layer interval 1.0mm, FOV50cm×50cm, the scanning time was 12s×5.

SUMMARY:
Fat infiltration and atrophy of lumbar muscles are related to spinal degenerative conditions, which can be seen reliably on MRI scans of lumbar disc herniation (LDH) patients. The aim of this study was to investigate the relationship between the degeneration of core muscles, obesity and chronic LDH. Fifty-five healthy volunteers and fifty-five chronic LDH patients (the course of the disease is more than six months) were enrolled. Core muscle percent fat and subcutaneous fat tissue thickness(SFTT) were used as the outcome measure, and logistic regression and independent samples t-test as the analytical methods to compare the relationship of the following five independent variables (erector spinae, rectus abdominis, [transversus abdominal, internal abdominal oblique, and external abdominal oblique muscle], lumbar multifidus, and psoas major muscles) and SFTT with LDH.

ELIGIBILITY:
Inclusion Criteria:

* patients in good physical health; ②patients aged 20 to 55 years, including 20 and 55 years, male or female; ③patients who agree to participate in the study and sign the informed consent.

Exclusion criteria:

* patients who performed lumbar and abdominal muscles exercises in the past; ②patients unable to tolerate magnetic resonance imaging or claustrophobia;

  * patients who are deemed unsuitable for the clinical trial.

Removing criteria:

* patients who decline participation of various reasons;

  * patients unable to comprehend questions asked by the researchers; ③patients intolerant to necessary examinations.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — patients and healthy volunteers aged 20 to 55 years, including 20 and 55 years
Study Population: Inclusion Criteria:
  ①patients who meet the diagnostic criteria for LDH based on overall consideration of their symptoms, signs, and radiological findings (MRI)； ②patients aged 20 to 55 years, including 20 and 55 years, male or female; ③Patients with a history of LDH for 6 months and/or above; ④patients who have signed the informed consent.
  Exclusion criteria:
  ①patients with LDH causing radiculopathy or cauda equina syndrome; ②patients with other diseases such as spinal stenosis, ankylosing spondylitis that causes low back pain; ③patients with a previous history of spinal surgery, traumatic injury to the spine; ④patients with bone tuberculosis, osteoporosis and bone tumors; ⑤patients with other severe cardiovascular and cerebrovascular diseases, digestive and hematopoietic system diseases; patients with diabetes mellitus Autoimmune diseases or other metabolic diseases; patients with mental diseases;
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
core muscles percent fat | baseline
  Magnetic resonance imaging-guided core muscles percent fat in patients with chronic LDH and healthy volunteers, including erector spinae, rectus abdominis, (transversus abdominal, internal abdominal oblique, and external abdominal oblique muscle), lumbar multifidus, and psoas major muscles was used as the outcome measure

SECONDARY OUTCOMES:
Subcutaneous fat tissue thickness | baseline
  Subcutaneous fat tissue thickness(SFTT) was measured as the vertical distance from the tip of spinous process to the skin on axial T2-weighted lumbar spine MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Shuguang Hospital Affiliated with Shanghai University of TCM, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes